CLINICAL TRIAL: NCT00598559
Title: A Phase III, Multi-Center, Open-Label, Prospective, Repeated Dose, Randomized, Controlled, Multi-Day Study of the Safety and Efficacy of Intravenous Acetaminophen in Adult Inpatients
Brief Title: Safety and Efficacy of Intravenous Acetaminophen (IV APAP) in Adult Inpatients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-APA-351
Record Dates: First submitted 2008-01-08; First posted 2008-01-22 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Acute Pain; Fever
Keywords: Acute pain; Fever; IV Acetaminophen; Analgesic
MeSH Terms: conditions — Acute Pain; Fever | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 g IV Acetaminophen (Experimental): 1 g q6h IV Acetaminophen
  Interventions: Drug: IV Acetaminophen
- 650 mg IV Acetaminophen (Experimental): 650 mg q4h IV Acetaminophen
  Interventions: Drug: IV Acetaminophen
- Standard of Care (Other): The standard of care treatments were defined as any medication the investigator deemed appropriate to treat the subject, including products containing acetaminophen but excluding IV acetaminophen.
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — Arm 1: 1 g IV Acetaminophen every 6 hours administered for five days. Arm 2: 650 mg IV Acetaminophen every 4 hours administered for five days. Arm 3: The standard of care treatments were defined as any medication the investigator deemed appropriate to treat the subject, including products containing acetaminophen but excluding IV acetaminophen.
  Other Names: IV Acetaminophen (IV APAP)

SUMMARY:
The study will be investigating safety and efficacy administration of repeated dose of IV Acetaminophen (IV APAP) over five days for the treatment of acute pain or fever in adult patients.

DETAILED DESCRIPTION:
• To assess the safety of IV Acetaminophen when used over five days for the treatment of acute pain or fever in adult inpatients

Secondary Objectives:

* To compare the efficacy of IV Acetaminophen 650 milligram (mg) every four (q4) hours vs. 1 gram (g) every 6 (q6) hours over 5 days of treatment
* To compare the safety of IV Acetaminophen 650 mg q4 hours vs. 1 g q6 hours over 5 days of treatment
* To compare the safety of IV Acetaminophen vs. standard of care (SOC) treatment over 5 days of treatment
* To compare the efficacy of IV Acetaminophen vs. standard of care treatment over 5 days of treatment

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participation in the Study
* Be at least 18 years of age and weigh at least 41 kilogram (kg)
* Be anticipated by the Investigator to require multi-day (target is five days) use of IV treatment either because of having a "nothing by mouth" (NPO) status having a medical condition that makes oral intake difficult having a medical condition that requires IV treatment
* Be willing to undergo 5 days of treatment with IV acetaminophen for the treatment of pain or fever (defined as a core temperature greater than or equal to 38 degrees celsius). Note that Subjects have a slightly less than 15% chance (one in seven) of being assigned to the Control Group and receiving standard of care treatment, but no IV APAP.
* Have the ability to read and understand the Study procedures and have the ability to communicate meaningfully with the Study Investigator and staff
* If a female of child bearing potential, have a negative pregnancy test within 48 hours of randomization

Exclusion Criteria:

* Has a significant medical disease, laboratory abnormality or condition that, in the Investigator's judgment, could compromise the Subject's welfare or would otherwise contraindicate Study participation
* Is expected to have difficulty in communicating with the Study staff or completing Study requirements (including follow up visits)
* Has known hypersensitivity to acetaminophen or the inactive ingredients (excipients) of IV acetaminophen or any contraindication to receiving acetaminophen
* Has impaired liver function, e.g., Alanine aminotransferase (ALT) greater than or equal to 3 times the upper limit of normal (ULN), bilirubin greater than or equal to 3 times ULN, known active hepatic disease (e.g., hepatitis), evidence of clinically significant chronic liver disease or other condition affecting the liver (e.g., alcoholism as defined by DSM-IV, cirrhosis or chronic hepatitis)
* Has participated in an interventional clinical Study (investigational or marketed product) within 30 days of Study entry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Viscusi, MD, Principal Investigator — Thomas Jefferson University
Locations (14):
- United States (14):
  - Arcadia Methodist Hospital, Arcadia, California
  - Glendale Adventist Medical Center, Glendale, California
  - Accurate Clinical Trials, Inc., Laguna Hills, California
  - Huntington Memorial Hospital, Pasadena, California
  - Lotus Clinical Research, Inc., Pasadena, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Nature Coast Clinical Research, Crystal River, Florida
  - G&G Research, Ft. Pierce, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Weill Medical College of Cornell University, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Memorial Herman/Memorial City Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open label study conducted in the US from 21 Feb 2008 -12 Aug 2008
Groups:
- IV Acetaminophen 1 Gram Every 6 Hours: All Subjects Randomized to Receive IV acetaminophen 1 gram administered every 6 hours.
- IV Acetaminophen 650 Milligram Every 4 Hours: All Subjects Randomized to Receive 650 mg IV acetaminophen administered every 4 hours.
- Standard of Care (SOC): All Subjects Randomized to Receive standard of care treatment under the discretion of the Investigator and the medical staff caring for them.
Period: Overall Study
Arm/Group | IV Acetaminophen 1 Gram Every 6 Hours | IV Acetaminophen 650 Milligram Every 4 Hours | Standard of Care (SOC)
Started | 92 | 91 | 30
Completed | 65 (Subjects completed 5 days of treatment) | 63 (Subjects completed 5 days of treatment) | 27 (Subjects completed 5 days of treatment)
Not Completed | 27 | 28 | 3
Not completed — Adverse Event | 11 | 7 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Protocol Non-compliance | 1 | 0 | 0
Not completed — Early discharge from hospital | 9 | 12 | 3
Not completed — Subject unable/unwilling to attend visit | 4 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- IV Acetaminophen 1g q6h: All Subjects Randomized to Receive IV acetaminophen 1g administered every 6 hours.
- IV Acetaminophen 650 mg q4h: All Subjects Randomized to Receive 650 mg IV acetaminophen administered every 4 hours.
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen 1g q6h | IV Acetaminophen 650 mg q4h | Standard of Care (SOC) | Total
Number analyzed (Participants) | 92 | 91 | 30 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 54 | 17 | 119
  >=65 years | 44 | 37 | 13 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 44 | 17 | 110
  Male | 43 | 47 | 13 | 103

OUTCOME MEASURES:

1. Secondary Outcome: Subject Global Evaluation of the Level of Satisfaction With Side Effects Related to Study Treatments
Description: Using a four point categorical scale 0= poor, 1= fair, 2= good, 3= excellent, comparisons of subject's Global Evaluations of the level of satisfaction with side effects related to study treatment at End of Day 5 (prior to discharge)
Time Frame: End of Day 5 (prior to discharge)
Population: Analyses were conducted using the mITT population, defined as subjects who were randomized to the IV acetaminophen groups and who received at least one dose of IV acetaminophen, and all subjects assigned to the SOC group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- IV Acetaminophen 1 g q6h: mITT Population, IV acetaminophen 1 g administered every 6 hours.
- IV Acetaminophen 650 mg q4h: mITT Population, IV acetaminophen 650 mg administered every 4 hours.
- Standard of Care (SOC): mITT Population, Subjects Who Received Standard of Care Treatment.
Arm/Group | IV Acetaminophen 1 g q6h | IV Acetaminophen 650 mg q4h | Standard of Care (SOC)
Number analyzed (Participants) | 64 | 63 | 26
Units on a scale | 2.5 (0.78) | 2.5 (0.67) | 2.0 (0.85)

2. Primary Outcome: Number of Subjects Reporting at Least One Treatment-Emergent Adverse Event (TEAE).
Description: Number of subjects who experienced at least one treatment emergent adverse event (TEAE).
  A TEAE is an adverse event that occurs on or after the first dose of study medication (T0).
Time Frame: T0 (first dose of IV APAP or randomization to SOC group) to Day 7 - 12 Follow-up
Population: Safety analyses were conducted using the mITT population, defined as subjects who were randomized to the IV acetaminophen groups and who received at least one dose of IV acetaminophen, and all subjects assigned to the SOC group.
Measure: Number; unit: Participants
Arm/Group | IV Acetaminophen 1 g q6h | IV Acetaminophen 650 mg q4h | Standard of Care (SOC)
Number analyzed (Participants) | 92 | 91 | 30
Participants | 77 | 86 | 26

3. Primary Outcome: Subjects Who Experienced at Least One Serious Treatment-Emergent Adverse Event (TEAE)
Description: Serious TEAE is any untoward medical occurrences at any dose of study medication that:
  * results in death
  * is life threatening
  * requires inpatient hospitalization or causes prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event
Time Frame: First dose (T0) to within 30 days of the last dose of study medication.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | IV Acetaminophen 1 g q6h | IV Acetaminophen 650 mg q4h | Standard of Care (SOC)
Number analyzed (Participants) | 92 | 91 | 30
Participants | 14 | 11 | 3

4. Secondary Outcome: Subject Global Evaluation of the Level of Satisfaction With Study Treatments Looking Back Over the Entire Treatment Period.
Description: Using a four point categorical scale 0= poor, 1= fair, 2= good, 3= excellent, comparisons of subject's Global Evaluations of the level of satisfaction with study treatments looking back over the entire treatment period was conducted at Day 7.
Time Frame: Study period lookback at Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | IV Acetaminophen 1 g q6h | IV Acetaminophen 650 mg q4h | Standard of Care (SOC)
Number analyzed (Participants) | 81 | 78 | 26
Units on a scale | 2.4 (0.75) | 2.3 (0.74) | 2.2 (0.61)

ADVERSE EVENTS:
Time Frame: AEs were collected after the start of study medication (T0) until approximately 7 days after the last dose for IVAPAP group or 12 days from T0 for SOC group. SAEs were collected from first dose until 30 days fter the last dose
Description: The end of the study date was:
  * IVAPAP:7 days from the last dose of study medication or maximum assessment date, whichever was greater.
  * SOC:12 days from T0 or maximum assessment date, whichever was greater.
Arm/Group | IV Acetaminophen 1 Gram Every 6 Hours | IV Acetaminophen 650 Milligram Every 4 Hours | Standard of Care (SOC)
Serious Adverse Events (participants affected / at risk) | 14/92 | 11/91 | 3/30
Other Adverse Events (participants affected / at risk) | 60/92 | 68/91 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen 1 Gram Every 6 Hours (N=92) | IV Acetaminophen 650 Milligram Every 4 Hours (N=91) | Standard of Care (SOC) (N=30)
Abscess (Infections and infestations) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 2 | 2 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Wound dehiscience (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen 1 Gram Every 6 Hours (N=92) | IV Acetaminophen 650 Milligram Every 4 Hours (N=91) | Standard of Care (SOC) (N=30)
Anaemia (Blood and lymphatic system disorders) | 11 | 10 | 6
Breath sounds abnormal (Investigations) | 7 | 6 | 1
Constipation (Gastrointestinal disorders) | 18 | 21 | 5
Headache (Nervous system disorders) | 7 | 5 | 4
Hypertension (Vascular disorders) | 6 | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 4 | 2
Hypotension (Vascular disorders) | 7 | 9 | 2
Insomnia (Psychiatric disorders) | 13 | 17 | 5
Nausea (Gastrointestinal disorders) | 23 | 34 | 8
Oedema peripheral (General disorders) | 7 | 7 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 13 | 2
Vomiting (Gastrointestinal disorders) | 6 | 10 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 2
Tachycardia (Cardiac disorders) | 5 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 1
Pyrexia (General disorders) | 4 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2 | 2
Anxiety (Psychiatric disorders) | 4 | 2 | 3
Phlebitis (Vascular disorders) | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
No separate efficacy analyses were performed for the fever because only 1 subject in each active group had fever as an indication, and no subject had both pain and fever as indications for treatment with IV acetaminophen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before any submission is made, Cadence shall be notified of the intention to publish and shall submit the manuscript to Cadence for review and comment.At least 60 days prior to submission for publication, investigator must submit manuscript to sponsor who has 60 days for review and comment. Publication may delayed at Cadence's written request for a period not to exceed 90 days if it contains a disclosure of an invention.